CLINICAL TRIAL: NCT04585698
Title: Quantitative Sensory Testing, Blink Reflex and Nociceptive Flexion Reflex in the Pathophysiology of Headache
Brief Title: QST, Blink Reflex and Nociceptive Flexion Reflex in Headache
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Manise Maite, Doctor in Medical Sciences, University of Liege
Other Study IDs: ULiege_CHEPS_AM_MM_JS
Record Dates: First submitted 2020-09-29; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Head Pain
Keywords: headache; fremanezumab; blink reflex; nociceptive flexion reflex; quantitative sensory testing
MeSH Terms: conditions — Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- headache patients
- healthy subjects

SUMMARY:
The aim of this study is to compare central and peripheric sensitization in headache patients at Baseline (T0) and 1 month after (T1) a treatment with an anti-CGRP (Fremanezumab-Ajovy).

DETAILED DESCRIPTION:
20 patients and 20 healthy subjects will be enrolled. The headache patients will be recruited just before starting their treatment and 1 month after (corresponding to the efficacy peak). Hot and cold stimulations will be delivered with the ATS probe from the Medoc Pathway on the forehead and on the hand (palmar face) to determine painful threshold to warm/cold stimuli. A blink reflex will be generated with a concentric electrode placed over the eyebrow and with active/earth electrodes linked to the EMG machine for the recording. For the nociceptive flexion reflex, a cutaneous stimulation will be applied on the arm and the response recorded on the corresponding muscles.

ELIGIBILITY:
Inclusion Criteria: patients with headache which are about to receive a treatment with fremanezumab

Exclusion Criteria:

* medication changes 1 month prior to the test
* neuropathy
* acute or chronic pain
* medications having effects on the central nervous system
* other disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with headache before and 1 month after receiving fremanezumab
  Age: 18-65 years
  Sex: 2/3 female, 1/3 male
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
modulation of pain threshold by fremanezumab | one year
  quantitative analysis of pain-related reflexes with QST (quantitative sensory testing) using Medoc Pathway
modulation of pain threshold by fremanezumab | one year
  Blink reflex and nociceptive flexion reflex usig EMG Viking Viasys.